CLINICAL TRIAL: NCT00825942
Title: An Open-Label Study of the Effect of C-KAD Ophthalmic Solution on Asteroid Hyalosis
Brief Title: An Open-Label Study of the Effect of an Ophthalmic Solution on Asteroid Hyalosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chakshu Research, Inc. (Industry)
Responsible Party: Ellen Hoogeveen /Associate Director, Clinical & Regulatory Affairs, Chakshu Research, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCK-0108
Record Dates: First submitted 2009-01-19; First posted 2009-01-21 (Estimated); Last update posted 2009-04-17 (Estimated); Status verified 2009-04

CONDITIONS: Asteroid Hyalosis
Keywords: Asteroid hyalosis; Opthalmic Study

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- C-KAD Ophthalmic Solution (Experimental)
  Interventions: Drug: C-KAD Ophthalmic Solution

INTERVENTIONS:
Drug: C-KAD Ophthalmic Solution — 4 drops applied daily for 180 days

SUMMARY:
To determine the safety and initial efficacy of C-KAD ophthalmic solution in patients with asteroid hyalosis

ELIGIBILITY:
Inclusion Criteria:

* Presence of asteroid hyalosis

Exclusion Criteria:

* Active ocular infection
* Glaucoma
* Ocular hypertension
* Ocular inflammatory disorders

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-10 (Estimated); Study Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
Reduction in the number of asteroid bodies | 180

CONTACTS AND LOCATIONS:
Overall Officials: Ira Wong, MD, Study Director — Chakshu Research, Inc.
Locations (1):
- Mountain View Optometry and Contact Lens Clinic, Mountain View, California, United States